CLINICAL TRIAL: NCT02893722
Title: A Randomized Double Blind Comparison of Atosiban in Patients With Repeated Implantation Failure Undergoing IVF Treatment
Brief Title: A Randomized Double Blind Comparison of Atosiban in Patients With RIF Undergoing IVF Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, chen zhi qin, associated clinical professor, Shanghai First Maternity and Infant Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FERRING-001
Record Dates: First submitted 2016-08-31; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Repeated Implantation Failure
Keywords: ivf ,atosiban,repeated implantation failure,RCT
MeSH Terms: interventions — atosiban; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- atosiban (Experimental): Give drugs 30 minutes before the start of the embryo transfer. First step: give a 37.5 mg Atosiban (Ferring, Germany) to take 0.9 ml, that is, 6.75 mg, conduct intravenous injection in one minute.
  Second step: for the remaining 4.1 ml, namely 30.75 mg, dilute to 41 ml, use the venous pump to adjust to 24 ml/h, infuse for 1 hour, namely 18 mg.
  Third step: for the remaining 17 ml, use the venous pump to adjust to 8 ml/h, infuse 2.1 hours, namely 12.75 mg. Total administration time is 3 hours, total dose is 37.5 mg.
  Interventions: Drug: atosiban
- 0.9% salain (Placebo Comparator): intravenous injection of 0.9% saline in one minute before transfer. Then use the same dose of normal saline for intravenous infusion to set the same infusion rate with experimental group, complete the infusion in 3 hours.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: atosiban — give drugs 30 minutes before the start of the embryo transfer,and intravenous infusion in total dose of 37.5 mg is set in certain infusion rate, and complete the infusion in 3 hours.
  Other Names: oxytocin antagonist
  Arms: atosiban
Drug: 0.9% saline — give drugs 30 minutes before the start of the embryo transfer,and intravenous infusion is set in the same rate with experimental group, complete the infusion in 3 hours.
  Other Names: Nacl
  Arms: 0.9% salain

SUMMARY:
This study intends to carry out a prospective, randomized, double blind and controlled study to compare the influence of Atosiban and placebo on uterine contraction frequency, endometrial blood flow perfusion, oxytocin and serum concentration of PGF2α, embryo implantation rate and clinical pregnancy rate on the RIF population after fresh embryo transfer, so as to further clarify the curative effect of Atosiban in the treatment of RIF and provide evidence-based basis for Atosiban for application in RIF population.

DETAILED DESCRIPTION:
Background and Rationale With the rapid development of the technology of reproductive medicine, in vitro fertilization embryo transfer (IVF-ET) and its related derivatives have become the most important means for the treatment of infertility. IVF-ET pregnancy rate increased from the initial 10% to current more than 50%, but the repeated implantation failure (RIF) has occurred occasionally, which has become a difficult that perplex IVF-ET clinical practices. There is no uniform definition of RIF at present. Coughlan et al called that the women below 40 years old who experienced at least 3 fresh or frozen periods and failed to transplant 4 and more than 4 high-quality embryos as RIF in 2014 [1]. At present, most of the patients have started the reason screening and inspection spontaneously if the transplantation fails after of transplanting 2 high-quality embryos. But the embryo implantation is a complex process, the etiology of RIF can be roughly summed as the embryo factors, uterine factors, genetic factors, immunological factors and so on, the symptomatic treatment according to different causes can improve the success rate of re-transplantation system [2]. However, in most cases, the etiology of RIF still cannot be explained [3].

In recent years, the influence of uterine contraction on embryo implantation has attracted more and more attention. Studies have shown that no matter it's natural menstrual cycle or fertility cycle, moderate Uterine Contraction (UC) is conducive to embryo implantation, but excessive or strong UC will have a negative impact on embryo implantation, and even the embryos to be implanted to the fallopian tube, cervical or vaginal, and even be discharged of the uterus [4-6].

The estrogen levels of excessively physiological state during the process of ovulation induction of IVF can induce the production ofoxytocin in the endometrial cells, and indirectly lead to the synthesis and release of prostaglandin PGF2α, resulting in increased uterine contraction frequency [7-9]. In 1998, Fanchin et al. found that the frequency of uterine contraction of about 30% of the embryos transplantation patients was higher than 5 times /min, which was significantly correlated to the success rate of low pregnancy [5]. The follow-up studies confirmed by ultrasound showed that the frequency of endometrial contraction induced by ovulation induction cycle of IVF[10] is 5-6 times of the natural cycle. Therefore, in addition to the soft operation of the transplant process, the reduction of uterine excessive contraction by drugs may be an effective measure to improve the success rate of IVF pregnancy.

Atosiban is the antagonist of mixed receptor of pitressin VIA and oxytocin, it competes the oxytocin receptor located on the uterine muscle cell membranes, foetal membrane and deciduas with oxytocin to inhibit contraction of the uterus; at the same time, it inhibits the generation of oxytocin induced uterine endometrial prostate element PGF2 α to increase the endometrial blood flow perfusion. Pierzynski et al first applied Atosiban to the field of reproduction in 2007 for the first time, which made the uterine contraction frequency of a RIF patient who failed to transplant for seven times before the oocyte donation embryo transplant decreased significantly, and successful became pregnant [11]. This report immediately caused the reproductive scientists to apply Atosiban to the clinical study of in vitro assisted reproduction. For the general population, there are still disputes on whether use Atosiban during the embryo transplant [12-14]. The prospective and randomized study of He Ye et al showed that Atosiban can significantly reduce the oxytocin of patients with endometriosis and serum concentrations of PGF2 α, reduce the frequency of uterine contraction and improve the implantation rate of quality blastocyst after freeze-thaw treatment and clinical pregnancy rate [15]. In the RIF population, the retrospective study and prospective cohort studies have shown that using low doses of Atosiban during IVF-ET can increase the implantation rate of fresh and thawed quality embryos and clinical pregnancy rate [16-18], which may improve pregnancy outcomes in patients with RIF. But these studies were not randomized placebo-controlled studies, and their conclusions are still to be verified.

Atosiban is currently a safe and effective tocolytic drug for uncomplicated preterm patients, the patients had accelerated heartbeat, nausea, vomiting, headache, dizziness, flushing, anxiety, tremor and other side effects occasionally. Randomized and double blind controlled trial showed that the side effects with application of Atosiban and placebo in the maternal and child was similar, the difference was not statistically significant [15]. Preclinical studies haven't found that Atosiban has any toxicity to human sperm motility or embryo development in rabbits [20]. It hasn't found the literatures that report the fetal congenital malformations associated with the application of Atosiban. Therefore, the therapeutic dose of Atosiban should be able to be safely used in embryo transfer.

In summary, this study intends to carry out a prospective, randomized, double blind and controlled study to compare the influence of Atosiban and placebo on uterine contraction frequency, endometrial blood flow perfusion, oxytocin and serum concentration of PGF2α, embryo implantation rate and clinical pregnancy rate on the RIF population after fresh embryo transfer, so as to further clarify the curative effect of Atosiban in the treatment of RIF and provide evidence-based basis for Atosiban for application in RIF population.

ELIGIBILITY:
Inclusion Criteria:

1. 3 or more than 3 embryo implantation failure histories previously (or the number of high-quality embryos transplanted is >4);
2. Age <40 years；
3. Ultrasound or HSG showed normal uterine cavity, endometrium on transplantation day is ≥ 8mm;
4. There's at least one good quality embryo on transplantation day.

Exclusion Criteria:

1. Patients using donor sperm or donor eggs;
2. Patients have obvious uterine cavity abnormalities;
3. There was a clear hydrosalpinx;
4. Natural cycles or IVM patients;
5. Patients who cancel the due to the transfer due to various reasons, such as the failure of fertilization, or ovarian transitional stimulus syndrome (OHSS);
6. Abnormal karyotype;
7. Blastocyst transplantation patients.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks after embryo transfer
  cases of clinical pregnancies / number of transplantation cycles(per patient)

SECONDARY OUTCOMES:
implantation rate | 4 weeks after embryo transfer
  number of pregnancy fetal bursa / total number of transplantation embryos
abortion rate | 6 weeks after embryo transfer
  abortion cases / number of clinical pregnancy cycles
ectopic pregnancy rate | 6 weeks after embryo transfer
  ectopic pregnancy cases / number of clinical pregnancy cycle
frequency of uterine contraction (4 minutes) | 1 hour before and 1 hour after intervention
  times of uterine contraction/4 minutes

OTHER OUTCOMES:
uterine artery blood flow index | 1 hour before and 1 hour after intervention
oxytocin and PGF2 α serum concentration. | 1 hour before and 1 hour after intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coughlan C, Ledger W, Wang Q, Liu F, Demirol A, Gurgan T, Cutting R, Ong K, Sallam H, Li TC. Recurrent implantation failure: definition and management. Reprod Biomed Online. 2014 Jan;28(1):14-38. doi: 10.1016/j.rbmo.2013.08.011. Epub 2013 Sep 14. PMID 24269084
- [Result] Simon A, Laufer N. Repeated implantation failure: clinical approach. Fertil Steril. 2012 May;97(5):1039-43. doi: 10.1016/j.fertnstert.2012.03.010. Epub 2012 Mar 30. PMID 22464086
- [Result] Margalioth EJ, Ben-Chetrit A, Gal M, Eldar-Geva T. Investigation and treatment of repeated implantation failure following IVF-ET. Hum Reprod. 2006 Dec;21(12):3036-43. doi: 10.1093/humrep/del305. Epub 2006 Aug 12. PMID 16905766
- [Result] Knutzen V, Stratton CJ, Sher G, McNamee PI, Huang TT, Soto-Albors C. Mock embryo transfer in early luteal phase, the cycle before in vitro fertilization and embryo transfer: a descriptive study. Fertil Steril. 1992 Jan;57(1):156-62. PMID 1730311
- [Result] Fanchin R, Righini C, Olivennes F, Taylor S, de Ziegler D, Frydman R. Uterine contractions at the time of embryo transfer alter pregnancy rates after in-vitro fertilization. Hum Reprod. 1998 Jul;13(7):1968-74. doi: 10.1093/humrep/13.7.1968. PMID 9740459
- [Result] Lesny P, Killick SR, Robinson J, Raven G, Maguiness SD. Junctional zone contractions and embryo transfer: is it safe to use a tenaculum? Hum Reprod. 1999 Sep;14(9):2367-70. doi: 10.1093/humrep/14.9.2367. PMID 10469712
- [Result] Richter ON, Kubler K, Schmolling J, Kupka M, Reinsberg J, Ulrich U, van der Ven H, Wardelmann E, van der Ven K. Oxytocin receptor gene expression of estrogen-stimulated human myometrium in extracorporeally perfused non-pregnant uteri. Mol Hum Reprod. 2004 May;10(5):339-46. doi: 10.1093/molehr/gah039. Epub 2004 Mar 25. PMID 15044599
- [Result] Liedman R, Hansson SR, Howe D, Igidbashian S, McLeod A, Russell RJ, Akerlund M. Reproductive hormones in plasma over the menstrual cycle in primary dysmenorrhea compared with healthy subjects. Gynecol Endocrinol. 2008 Sep;24(9):508-13. doi: 10.1080/09513590802306218. PMID 18958771
- [Result] Zhu L, Li Y, Xu A. Influence of controlled ovarian hyperstimulation on uterine peristalsis in infertile women. Hum Reprod. 2012 Sep;27(9):2684-9. doi: 10.1093/humrep/des257. Epub 2012 Jul 14. PMID 22798632
- [Result] Ayoubi JM, Epiney M, Brioschi PA, Fanchin R, Chardonnens D, de Ziegler D. Comparison of changes in uterine contraction frequency after ovulation in the menstrual cycle and in in vitro fertilization cycles. Fertil Steril. 2003 May;79(5):1101-5. doi: 10.1016/s0015-0282(03)00179-1. PMID 12738502
- [Result] Pierzynski P, Reinheimer TM, Kuczynski W. Oxytocin antagonists may improve infertility treatment. Fertil Steril. 2007 Jul;88(1):213.e19-22. doi: 10.1016/j.fertnstert.2006.09.017. Epub 2007 May 3. PMID 17481622
- [Result] Moraloglu O, Tonguc E, Var T, Zeyrek T, Batioglu S. Treatment with oxytocin antagonists before embryo transfer may increase implantation rates after IVF. Reprod Biomed Online. 2010 Sep;21(3):338-43. doi: 10.1016/j.rbmo.2010.04.009. Epub 2010 Apr 18. PMID 20638340
- [Result] Song XR, Zhao XH, Bai XH, Lu YH, Zhang HJ, Wang YX, Lu R. [Application of oxytocin antagonists in thaw embryo transfer]. Zhonghua Fu Chan Ke Za Zhi. 2013 Sep;48(9):667-70. Chinese. PMID 24332133
- [Result] Ng EH, Li RH, Chen L, Lan VT, Tuong HM, Quan S. A randomized double blind comparison of atosiban in patients undergoing IVF treatment. Hum Reprod. 2014 Dec;29(12):2687-94. doi: 10.1093/humrep/deu263. Epub 2014 Oct 21. PMID 25336707
- [Result] He Y, Wu H, He X, Xing Q, Zhou P, Cao Y, Wei Z. Administration of atosiban in patients with endometriosis undergoing frozen-thawed embryo transfer: a prospective, randomized study. Fertil Steril. 2016 Aug;106(2):416-22. doi: 10.1016/j.fertnstert.2016.04.019. Epub 2016 Apr 30. PMID 27143518
- [Result] Lan VT, Khang VN, Nhu GH, Tuong HM. Atosiban improves implantation and pregnancy rates in patients with repeated implantation failure. Reprod Biomed Online. 2012 Sep;25(3):254-60. doi: 10.1016/j.rbmo.2012.05.014. Epub 2012 Jun 16. PMID 22818095
- [Result] Chou PY, Wu MH, Pan HA, Hung KH, Chang FM. Use of an oxytocin antagonist in in vitro fertilization-embryo transfer for women with repeated implantation failure: a retrospective study. Taiwan J Obstet Gynecol. 2011 Jun;50(2):136-40. doi: 10.1016/j.tjog.2011.04.003. PMID 21791296
- [Result] Zhang Yue, Zhu Yujing, Luo Haining, et al. Clinical observation on the effect of the patients using Atosiban for frozen thawed embryo transfer after repeated failure of implantation. Chinese Journal of Family Planning,2016,22 (05): 325-328.
- [Result] Romero R, Sibai BM, Sanchez-Ramos L, Valenzuela GJ, Veille JC, Tabor B, Perry KG, Varner M, Goodwin TM, Lane R, Smith J, Shangold G, Creasy GW. An oxytocin receptor antagonist (atosiban) in the treatment of preterm labor: a randomized, double-blind, placebo-controlled trial with tocolytic rescue. Am J Obstet Gynecol. 2000 May;182(5):1173-83. doi: 10.1067/mob.2000.95834. PMID 10819855
- [Result] Pierzynski P, Gajda B, Smorag Z, Rasmussen AD, Kuczynski W. Effect of atosiban on rabbit embryo development and human sperm motility. Fertil Steril. 2007 May;87(5):1147-52. doi: 10.1016/j.fertnstert.2006.08.089. Epub 2007 Jan 16. PMID 17224148
- [Derived] Tang CL, Li QY, Chen FL, Cai CT, Dong YY, Wu YY, Yang JZ, Zhao M, Chi FL, Hong L, Ai A, Chen MX, Li KM, Teng XM, Chen ZQ. A randomized double blind comparison of atosiban in patients with recurrent implantation failure undergoing IVF treatment. Reprod Biol Endocrinol. 2022 Aug 19;20(1):124. doi: 10.1186/s12958-022-00999-y. PMID 35986323
- [Derived] Craciunas L, Tsampras N, Kollmann M, Raine-Fenning N, Choudhary M. Oxytocin antagonists for assisted reproduction. Cochrane Database Syst Rev. 2021 Sep 1;9(9):CD012375. doi: 10.1002/14651858.CD012375.pub2. PMID 34467530